CLINICAL TRIAL: NCT04487210
Title: A Phase I, Prospective, Open-Labeled Study to Evaluate the Safety and Immunogenicity of MVC-COV1901
Brief Title: A Study to Evaluate the Safety and Immunogenicity of MVC-COV1901 Against COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CT-COV-11
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
Keywords: COVID-19 vaccine
MeSH Terms: conditions — COVID-19 | interventions — MVC-COV1901 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1a (Low Dose) (Experimental): 15 subjects will be enrolled to receive Low-dose S-protein with adjuvant MVC-COV1901.
  Interventions: Biological: MVC-COV1901
- Phase 1b (Medium Dose) (Experimental): 15 subjects will be enrolled to receive Medium-dose S-protein with adjuvant MVC-COV1901.
  Interventions: Biological: MVC-COV1901
- Phase 1c (High Dose) (Experimental): 15 subjects will be enrolled to receive High-dose S-protein with adjuvant MVC-COV1901.
  Interventions: Biological: MVC-COV1901

INTERVENTIONS:
Biological: MVC-COV1901 — MVC-COV1901 is formulated in the different dosages of Spike (S) protein with CpG 1018 and aluminum content as adjuvant.

SUMMARY:
This is a phase I prospective, open-labeled, single-center study to evaluate the safety and immunogenicity of MVC-COV1901.

DETAILED DESCRIPTION:
This is a phase I prospective, open-labeled, single-center study to evaluate the safety and immunogenicity of MVC-COV1901. This study is a dose escalation study with three separate arms for subjects at the age of ≥20 and <50 years. The vaccination schedule for primary regimen consists of two doses of MVC-COV1901 for each study subject, administered by intramuscular (IM) injection 0.5mL in the deltoid region of non-dominant arm preferably 28 days apart, on Day 1 and Day 29. Subjects will receive a single booster vaccination of MVC-COV1901 on Day 209, 180 days after completion of the primary regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy volunteer ≥20 and <50 years of age
2. Subject free of ongoing acute diseases or serious medical conditions (e.g. concomitant illness) such as cardiovascular (e.g. New York Heart Association grade III or IV), hepatic (e.g. Child-Pugh Class C), psychiatric condition (e.g. alcoholism, drug abuse), medical history, physical findings, or laboratory abnormality that in the investigator's opinion could interfere with the results of the trial or adversely affect the safety of the subject
3. Female subject must be:

   * Either of non-childbearing potential, i.e. surgically sterilized (defined as having undergone hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year post-menopausal;
   * Or, if of childbearing potential, must be abstinent or agree to use medically effective contraception from 14 days before screening to 30 days following last injection of study vaccines. Acceptable forms include:
   * Implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS)
   * Established use of hormonal methods (injectable, pill, patch or ring) combined with barrier methods of contraception: condom, or occlusive cap (diaphragm or cervical/vault caps) withspermicidal foam/gel/film/cream/suppository
   * Have a negative pregnancy test
4. Subject is willing and able to comply with all required study visits and follow-up required by this protocol
5. Subject has no overseas travel within 14 days of screening and will not have any throughout the study period
6. Subject must provide written informed consent or the Subject's legal representative must understand and consent to the procedure

Exclusion Criteria:

1. Receiving any investigational intervention either currently or within 30 days of first dose;
2. Subject (particularly who is a healthcare worker) with previous known or potential exposure to SARS CoV-1 or 2 viruses (EXCEPT for those who have been tested negative and the 14-days self-managements/ home quarantines/ home isolations are completed), or received any other COVID-19 vaccine;
3. Administration of any vaccine within 4 weeks of first dose;
4. A BMI greater than or equal to 30 kg/m2;
5. Subject with a history of hypersensitivity to any vaccine or a history of allergic disease or reactions likely to be exacerbated by any component of the MVC-COV1901;
6. Administration of any blood product or intravenous immunoglobulin administration within 12 weeks of first dose;
7. Pregnancy or breast feeding or have plans to become pregnant in 30 days after last injection of study vaccines;
8. History of positive serologic test for HIV, hepatitis B surface antigen (HBsAg) or any potentially communicable infectious disease as determined by the investigator or Medical Monitor;
9. Positive serologic test for hepatitis C (EXCEPTION: successful treatment with confirmation of sustained virologic response);
10. Baseline evidence of kidney disease as measured by creatinine greater than 1.5 mg/dL;
11. Screening laboratory tests with Grade 2 or higher abnormality (Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, September 2007);
12. Immunosuppressive illness including hematologic malignancy, history of solid organ or bone marrow transplantation;
13. A history of autoimmune disease (systemic lupus, rheumatoid arthritis, scleroderma, polyarthritis, thyroiditis, etc.);
14. Current or anticipated concomitant immunosuppressive therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or less than prednisone 20 mg/day or equivalent) within 12 weeks of first dose;
15. Current or anticipated treatment with TNF-α inhibitors, e.g. infliximab, adalimumab, etanercept within 12 weeks of first dose;
16. Prior major surgery or any radiation therapy within 12 weeks of first dose;
17. Alcohol or drug abuse or dependence, psychiatric, addictive, or any disorder that, in the opinion of the investigator, would interfere with adherence to study requirements or assessment of immunologic endpoints; or any illness or condition that in the opinion of the investigator may affect the safety of the participant or the evaluation of any study endpoint;
18. Presence of keloid scar formation or hypertrophic scar as a clinically significant medical condition, tattoos or wound covering the injection site area;
19. Body (oral, rectal or ear) temperature ≥ 38.0°C or acute illness within 2 days of first dose, or acute respiratory illness within 14 days of first dose;
20. Screening laboratory test of antinuclear antibody (ANA), anti-dsDNA antibody, anti-neutrophil cytoplasmic antibodies (ANCA, including cytoplasmic ANCA (c-ANCA), perinuclear ANCA (p-ANCA)) with the value higher than upper normal limit;
21. Abnormal screening electrocardiography (ECG) with clinically significant findings as reviewed by investigator.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Safety of MVC-COV1901 | Day 1 to 28 days after second vaccination
  Incidence of solicited adverse events (AEs) after vaccination, Incidence of unsolicited AEs and other AEs after vaccination, Incidence of laboratory abnormality after vaccination, Incidence of adverse event of special interest (AESI) and serious adverse events (SAEs) after vaccination

SECONDARY OUTCOMES:
Immunogenicity (neutralizing antibody titers and antigen specific binding antibody titers) | 14 days, 28 days after each vaccination, and 180 days after second vaccination.
  Geometric mean titer (GMT)
Immunogenicity (neutralizing antibody titers and antigen specific binding antibody titers) | 14 days, 28 days after each vaccination, and 180 days after second vaccination.
  Seroconversion rate (SCR)
Immunogenicity (neutralizing antibody titers and antigen specific binding antibody titers) | 14 days, 28 days after each vaccination, and 180 days after second vaccination.
  GMT ratio
Immunogenicity (antigen specific cellular immune responses) | 28 days and 180 days after second vaccination
  The positive rate of cellular mediated immune response
Safety of MVC-COV1901 | Day 1 to Day 209
  Incidence of other adverse events, Incidence of adverse event of special interest (AESI) and serious adverse events (SAEs) within the study period
Immunogenicity (neutralizing antibody titers and antigen specific binding antibody titers) | 28 days and 180 days after the booster vaccination.
  Geometric mean titer (GMT)
Immunogenicity (neutralizing antibody titers and antigen specific binding antibody titers) | 28 days and 180 days after the booster vaccination.
  Seroconversion rate (SCR)
Immunogenicity (neutralizing antibody titers and antigen specific binding antibody titers) | 28 days and 180 days after the booster vaccination.
  GMT ratio

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hsieh SM, Chang SC, Cheng HY, Shih SR, Lien CE. Durability and Immunogenicity of Neutralizing Antibodies Response Against Omicron Variants After Three Doses of Subunit SARS-CoV-2 Vaccine MVC-COV1901: An Extension to an Open-Label, Dose-Escalation Phase 1 Study. Infect Dis Ther. 2022 Aug;11(4):1493-1504. doi: 10.1007/s40121-022-00652-6. Epub 2022 May 17. PMID 35579840
- [Derived] Hsieh SM, Liu WD, Huang YS, Lin YJ, Hsieh EF, Lian WC, Chen C, Janssen R, Shih SR, Huang CG, Tai IC, Chang SC. Safety and immunogenicity of a Recombinant Stabilized Prefusion SARS-CoV-2 Spike Protein Vaccine (MVC-COV1901) Adjuvanted with CpG 1018 and Aluminum Hydroxide in healthy adults: A Phase 1, dose-escalation study. EClinicalMedicine. 2021 Aug;38:100989. doi: 10.1016/j.eclinm.2021.100989. Epub 2021 Jun 26. PMID 34222848